CLINICAL TRIAL: NCT03554902
Title: Endoscopic Gastric Tubulization
Acronym: Endosleeve
Status: Recruiting | Type: Observational
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Other Study IDs: 16-001-OBS (CPP); 2017-A03599-44 (Other: ANSM France)
Record Dates: First submitted 2018-05-16; First posted 2018-06-13 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Morbid Obesity
Keywords: Endoscopic gastric tubulization; Weight loss; Quality of life
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Endoscopic gastric tubulization: Endoscopic gastric tubulization is performed using the CE marked endoscopic suture device Overstitch (Apollo Endosurgery, Austin, Tx. USA).
  Interventions: Procedure: Endoscopic gastric tubulization

INTERVENTIONS:
Procedure: Endoscopic gastric tubulization — Endoscopic gastric tubulization is performed using the CE marked endoscopic suture device Overstitch (Apollo Endosurgery, Austin, Tx. USA).

SUMMARY:
Endoscopic gastric tubulization is currently proposed in the Digestive Surgery Department of the Nouvel Hôpital Civil, Strasbourg, France, to adult patients with morbid obesity. The procedure is performed using the CE marked endoscopic suture device Overstitch (Apollo Endosurgery, Austin, Tx. USA). It is standard practice since October 2016.

The objective of this study is to prospectively collect data of patients who underwent an endoscopic gastric tubulization, from last visit before procedure to 2 years after procedure. These data are usually collected during medical consultations and will enable the evaluation of weight loss, quality of life and comorbidities improvement, reproducibility and durability of the technique.

DETAILED DESCRIPTION:
Gastric restriction is one of the fundamental principles of gastric bypass and gastric banding. Despite its advantages (long term weight loss, comorbidities related to obesity improvement…), bariatric surgery is risky. In fact, complications putting the patient into a life-threatening condition can occur. Endoscopic approaches are similar to current surgical methods but less invasive, safer and allow ambulatory care.

Nowadays, practitioners have the possibility to reduce stomach size by merging tissues through an endoscopic endoluminal suture approach without any incision. This leads to similar results (gastric restriction, weight loss, quality of life and comorbidities improvement) compared with standard surgical procedure while reducing the risk of complications.

One of the major benefit of this technique is its reversibility. A new surgical or endoscopic procedure is possible at a later stage.

Endoscopic gastric tubulization is currently proposed in the Digestive Surgery Department of the Nouvel Hôpital Civil, Strasbourg, France, to adult patients with morbid obesity. The procedure is performed using the CE marked endoscopic suture device Overstitch (Apollo Endosurgery, Austin, Tx. USA). It is standard practice since October 2016.

The objective of this study is to prospectively collect data of patients who underwent an endoscopic gastric tubulization, from last visit before procedure to 2 years after procedure. These data are usually collected during medical consultations and will enable the evaluation of weight loss, quality of life and comorbidities improvement, reproducibility and durability of the technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an endoscopic gastric tubulization in the Nouvel Hôpital Civil, Strasbourg, France

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old requiring a treatment for morbid obesity.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-06-08 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in weight loss | 7 days, 1 - 3 - 6 - 9 - 12 - 18 and 24 months after procedure
  Change in weight loss measured in kilograms.
Change in excess weight loss | 7 days, 1 - 3 - 6 - 9 - 12 - 18 and 24 months after procedure
  Change in excess weight loss measured in percentage. Excess weight loss = (weight loss at time point / weight loss goal to reach a body mass index of 25 kg/m²) x 100
Change in body mass index variation | 7 days, 1 - 3 - 6 - 9 - 12 - 18 and 24 months after procedure
  Change in body mass index variation measured in kg/m².

SECONDARY OUTCOMES:
Number of patients with procedure-related adverse event | 7 days, 1 - 3 - 6 - 9 and 12 months after procedure
  Number of patients with procedure-related adverse event within 12 months after procedure.
Comorbidities improvement | 7 days, 1 - 3 - 6 - 9 - 12 - 18 and 24 months after procedure
  Improvement of sleep apnea, arterial hypertension, diabetes, reflux, osteoarticular disorders compared with preoperative data.
Quality of life improvement | 3 - 12 - 18 and 24 months after procedure
  Improvement of quality of life assessed by Moorehead-Ardelt Quality of Life questionnaire II. Score range from -3.0 to 3.0.
  * Score from -3.0 to -2.1: very poor quality of life
  * Score from -2.0 to -1.1: poor quality of life
  * Score from -1.0 to 1.0: fair quality of life
  * Score from 1.1 to 2.0: good quality of life
  * Score from 2.1 to 3.0: very good quality of life.
Gastro-intestinal quality of life improvement | 3 - 12 - 18 and 24 months after procedure
  Improvement of quality of life assessed by the Gastro-Intestinal Quality of Life Index questionnaire. A global score > 125 is considered as normal.
Modification in the feeling of satiety | 1 - 3 - 6 - 12 - 18 and 24 months after procedure
  Satiety assessed by Three Factors Eating Questionnaire - R18. Three dimensions are assessed. The higher the score is, the more important the dimension is.
  * Restrained eating: score from 6 to 24
  * Uncontrolled eating: score from 9 to 36
  * Emotional eating: score from 3 to 12.
Upper GI tract radiologic evaluation | 1 day, 6 - 12 and 24 months after procedure
  Upper GI control series.
Upper GI tract endoscopic evaluation | 6 - 12 and 24 months after procedure
  Upper GI control gastroscopy.
Procedure duration | At time of procedure
  Time required to perform the endoscopic gastric tubulization.
Number of stitches in place | At time of procedure
  Number of stitches put in place during the endoscopic gastric tubulization.

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Perretta, MD, PhD, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil - Strasbourg; Michel Vix, MD, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil - Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez-Nava G, Galvao MP, da Bautista-Castano I, Jimenez A, De Grado T, Fernandez-Corbelle JP. Endoscopic sleeve gastroplasty for the treatment of obesity. Endoscopy. 2015 May;47(5):449-52. doi: 10.1055/s-0034-1390766. Epub 2014 Nov 7. PMID 25380508
- [Background] Lopez-Nava G, Galvao MP, Bautista-Castano I, Jimenez-Banos A, Fernandez-Corbelle JP. Endoscopic Sleeve Gastroplasty: How I Do It? Obes Surg. 2015 Aug;25(8):1534-8. doi: 10.1007/s11695-015-1714-7. PMID 26003549
- [Background] Lopez-Nava G, Galvao M, Bautista-Castano I, Fernandez-Corbelle JP, Trell M. Endoscopic sleeve gastroplasty with 1-year follow-up: factors predictive of success. Endosc Int Open. 2016 Feb;4(2):E222-7. doi: 10.1055/s-0041-110771. Epub 2016 Jan 15. PMID 26878054
- [Background] Sharaiha RZ, Kedia P, Kumta N, DeFilippis EM, Gaidhane M, Shukla A, Aronne LJ, Kahaleh M. Initial experience with endoscopic sleeve gastroplasty: technical success and reproducibility in the bariatric population. Endoscopy. 2015 Feb;47(2):164-6. doi: 10.1055/s-0034-1390773. Epub 2014 Nov 7. PMID 25380510
- [Background] Abu Dayyeh BK, Rajan E, Gostout CJ. Endoscopic sleeve gastroplasty: a potential endoscopic alternative to surgical sleeve gastrectomy for treatment of obesity. Gastrointest Endosc. 2013 Sep;78(3):530-5. doi: 10.1016/j.gie.2013.04.197. Epub 2013 May 24. PMID 23711556